CLINICAL TRIAL: NCT02900404
Title: VeriXAPPORT: Verification of XAPPORT: a Decision Support App for Physicians Used for Patients Anticoagulated With Rivaroxaban in Terms of Anticoagulation Management in Elective Surgery: Verification Process of Medical Decision Algorithm
Brief Title: Verification of XAPPORT: a Decision Support App for Physicians Used for Patients Anticoagulated With Rivaroxaban in Terms of Anticoagulation Management in Elective Surgery: Verification Process of Medical Decision Algorithm
Acronym: VeriXAPPORT
Status: Withdrawn | Type: Observational
Why Stopped: due to release of competing App
Sponsor: Bayer (Industry)
Collaborators: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 18903
Record Dates: First submitted 2016-08-22; First posted 2016-09-14 (Estimated); Last update posted 2024-11-13 (Actual); Status verified 2017-04

CONDITIONS: Atrial Fibrillation; Venous Thromboembolism; Pulmonary Embolism
MeSH Terms: conditions — Atrial Fibrillation; Venous Thromboembolism; Pulmonary Embolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- NVAF Patients: Adult female and male patients with non-valvular atrial fibrillation (NVAF) treated with rivaroxaban before and after surgery
  Interventions: Other: XAPPORT; Other: Expert Panel ("gold standard")
- VTE/PE Patients: Adult female and male patients with venous thromboembolism/pulmonary embolism (VTE/PE) treated with rivaroxaban before and after surgery
  Interventions: Other: XAPPORT; Other: Expert Panel ("gold standard")

INTERVENTIONS:
Other: XAPPORT — A mobile device app based on different guidelines provides adequate guidance to physicians attending patients undergoing elective surgery, who have to interrupt treatment with rivaroxaban for surgery, in deciding how to approach the pre- and postoperative management of anticoagulation.
Other: Expert Panel ("gold standard") — A national panel of experts comprising anesthetists and surgeons from various disciplines advised in developing an algorithm supporting physicians how to approach the perioperative management of anticoagulation in patients receiving rivaroxaban and requiring elective surgery.

SUMMARY:
This study shall determine whether XAPPORT - a mobile device app based on different guidelines, the summary of product characteristics of rivaroxaban, and clinical facts and practice - provides adequate guidance to physicians attending patients undergoing elective surgery, who have to interrupt treatment with rivaroxaban for surgery, in deciding how to approach the pre- and postoperative management of anticoagulation.

DETAILED DESCRIPTION:
Study design: "retrospective/prospective" Observational study

ELIGIBILITY:
Inclusion Criteria:

* Female or male patient ≥18 years who provided signed and dated informed consent to the use of their medical data
* Patient was treated with rivaroxaban before and after surgery because of non-valvular atrial fibrillation (NVAF) or venous thromboembolism/pulmonary embolism (VTE/PE)
* Elective surgery in a department of General Surgery or Orthopedics / Trauma Surgery was performed within the last 12 months before study start
* The patient has been discharged from hospital
* Patient's medical records are available for data entry

Exclusion Criteria:

* Patient participated in an interventional drug study within 3 months prior to the surgery and discharge from hospital

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: At least 100 evaluable female or male inpatients shall be enrolled after having been discharged from hospital and provide data for analyses. Patients meeting all inclusion criteria and no exclusion criterion are suitable for this study. Enrolment will continue until at least 100 patients with complete data for analysis are available (i.e. 100 evaluable patients). An adequate representation of every bleeding and thromboembolism risk category per indication in the matrix will be taken into account.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-02-15 (Estimated); Primary Completion 2017-03-31 (Estimated); Study Completion 2017-03-31 (Estimated)

PRIMARY OUTCOMES:
Agreement rate between the recommendations of XAPPORT and the consolidated recommendations of a qualified Expert Panel ("gold standard"). | 4 months

SECONDARY OUTCOMES:
Reasons for discrepancies between the recommendations of XAPPORT and the consolidated recommendations of the qualified Expert Panel ("gold standard"). | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer